CLINICAL TRIAL: NCT05752032
Title: A Long Term Follow-up Study of Subjects Who Received ICM-203 or Matching Placebo
Status: Enrolling by invitation | Type: Observational
Sponsor: ICM Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICM 20-1002
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Adeno-associated virus; Gene therapy; ICM-203; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICM-203: Participants who previously received ICM-203 in ICM-203 clinical studies
  Interventions: Genetic: ICM-203
- Placebo: Participants who previously received placebo in ICM-203 clinical studies
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: ICM-203 — Long term follow-up
  Groups: ICM-203
Drug: Placebo — Long term follow-up
  Groups: Placebo

SUMMARY:
This is an observational study of the long term safety and efficacy of ICM-203.

DETAILED DESCRIPTION:
Subjects who have received ICM-203 or matching placebo from ICM-203 clinical studies will be enrolled. Subjects will be contacted annually to collect safety and efficacy outcomes until 5 years after the last dose of ICM-203 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Previous receipt of ICM-203 or matching placebo

Exclusion Criteria:

* None

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who received ICM-203 or matching placebo in clinical studies
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed adverse events | Up to 5 years

SECONDARY OUTCOMES:
Knee pain | Up to 3 years
  Evaluation of change from baseline in knee pain as measured using a Numerical Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable)
Knee function | Up to 3 years
  Evaluation of change from baseline in knee function as measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS) function in daily living subscale ranging from 0 (extreme problems) to 100 (no problems)
Magnetic Resonance Imaging Osteoarthritis Knee Score (MOAKS) | Up to 3 years
  Evaluation of change from baseline in MOAKS, focusing on bone marrow lesions, articular cartilage, and effusion-synovitis, where higher scores reflect worse disease
Joint space width | Up to 3 years
  Evaluation of change from baseline in joint space width in mm as measured on knee radiograph
Incidence of total knee replacement | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alison Heald, MD, Study Director — ICM Co. Ltd.
Locations (2):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Barwon Health, Geelong, Victoria

IPD SHARING:
Plan to Share IPD: No